CLINICAL TRIAL: NCT03115645
Title: Evaluation of the Dynamic Work Intervention for Office Workers to Reduce Sedentary Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Achmea (Other)
Responsible Party: Principal Investigator, H. P. Van der Ploeg, Associate Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DynamicWork
Record Dates: First submitted 2017-02-08; First posted 2017-04-14 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Lifestyle-related Condition
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive the Dynamic Working Intervention program, as described in the next section.
  Interventions: Other: Dynamic Work
- Control group (No Intervention): Participants in the control group will not receive any intervention and will perform their work in the same manner as before.

INTERVENTIONS:
Other: Dynamic Work — The intervention consists of the introduction of sit-stand workstations and desk bikes in the participants work environment in a ratio of 1:2 with traditional desks and chairs. Employees will receive a half hour intervention session at the start of the intervention from an occupational physiotherapist, who will provide further intervention support in the ensuing 12 weeks. Intervention participants will also receive an activity tracker which provides feedback on sitting time and physical activity levels.
  Other Names: Dynamisch Werken
  Arms: Intervention group

SUMMARY:
Long-term sitting has been associated with multiple health risks. To reduce sitting time for office workers in a Dutch insurance company, an intervention will be implemented. The goal of this study is to evaluate this intervention on the short term (3 months) and long-term (12 months).

DETAILED DESCRIPTION:
Large volumes of sitting time have been associated with multiple health risks such as diabetes, heart disease and premature death. Especially, in office workers sitting time per day can accumulate to over 10 hours a day. To reduce sitting time for office workers in a Dutch insurance company, an intervention will be implemented. The intervention contains the introduction of alternative workstations, intervention sessions with an occupational physiotherapist and an activity tracker with a self-help program booklet. The goal of this study is to evaluate the (cost) effectiveness of this intervention on the short term (3 months) and long-term (12 months). The primary outcome is objectively assessed sitting time.

In a cluster randomized controlled trial 250 employees of an insurance company will participate in the study. After baseline measurements, matched departments will be randomly assigned to the control or intervention group. The evaluation includes an economic and process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Employed by the insurance company for at least the duration of the study (12 months)
* Employed at least 28 hours per week
* Employed at one of the participating departments

Exclusion Criteria:

* Already access to the Dynamic Working Intervention
* Unable to stand or walk for longer time periods (i.e. wheelchair bound)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Sitting time | Change in sitting time between baseline and 12 month follow up assessment
  Total sitting time will be measured objectively with the activPAL activity tracker

SECONDARY OUTCOMES:
Occupational sitting time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, occupational time will be recorded and linked with a diary
Non-occupational sitting time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, non-occupational time will be recorded and linked with a diary
Total standing time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker
Occupational standing time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, occupational time will be recorded and linked with a diary
Non-occupational standing time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, non-occupational time will be recorded and linked with a diary
Total stepping time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker
Occupational stepping time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, occupational time will be recorded and linked with a diary
Non-occupational stepping time | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, non-occupational time will be recorded and linked with a diary
Sitting time in bouts of 30 min | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker
Occupational sitting time in bouts of 30 min | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, occupational time will be recorded and linked with a diary
Non-occupational sitting time in bouts of 30 min | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, non-occupational time will be recorded and linked with a diary
Sitting time in bouts of 60 min | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker
Occupational sitting time in bouts of 60 min | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, occupational time will be recorded and linked with a diary
Non-occupational sitting time in bouts of 60 min | Assessed at baseline 3 months and 12 months
  Objectively assessed by the activPAL activity tracker, non-occupational time will be recorded and linked with a diary
Waist circumference and body height | Assessed at baseline 3 months and 12 months
  Waist circumference and body height will be objectively measured in cm
Body weight | Assessed at baseline 3 months and 12 months
  Body weight will be objectively measured in kg and used to calculate body mass index (BMI)
Individual Work Performance | Assessed at baseline 3 months and 12 months
  Will be assessed with the Individual Work Performance Questionnaire (IWPQ)
Need for recovery | Assessed at baseline 3 months and 12 months
  This will be assessed with the Need For Recovery (NFR) questionnaire
Effort-reward imbalance | Assessed at baseline 3 months and 12 months
  This will be assessed with the short Effort-Reward Imbalance (ERI-short) questionnaire
Musculoskeletal complaints | Assessed at baseline 3 months and 12 months
  This will be assessed with the Nordic Musculoskeletal questionnaire
Vitality | Assessed at baseline 3 months and 12 months
  This will be assessed with the Vita-16© TNO questionnaire
Quality of life measured with EQ-5D-5L | Assessed at baseline 3 months and 12 months
  This will be assessed with the EQ-5D-5L questionnaire
Absenteeism | Assessed at baseline 3 months and 12 months
  This will be self-reported as well as assessed with company records
Healthcare consumption | Assessed at 3 months and 12 months
  This includes general practitioner, allied health professionals, complementary medicine consumption
Sitting, physical activity and work related outcomes | Assessed at baseline 3 months and 12 months
  These will be assessed with custom sitting, physical activity and work questions
Process evaluation | Assessed at 3 months and 12 months
  A process evaluation will be performed using qualitative (focus group interviews) and quantitative methods (questionnaires) in order to determine the level of implementation of the intervention as well as barriers and facilitators of this implementation.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Achmea, Apeldoorn
  - Achmea, Leeuwarden
  - Achmea, Leusden
  - Achmea, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jelsma JGM, van der Ploeg HP, Renaud LR, Stijnman DPM, Loyen A, Huysmans MA, van der Beek AJ, van Nassau F. Mixed-methods process evaluation of the Dynamic Work study: A multicomponent intervention for office workers to reduce sitting time. Appl Ergon. 2022 Oct;104:103823. doi: 10.1016/j.apergo.2022.103823. Epub 2022 Jun 17. PMID 35724470
- [Derived] Mastenbroek VJEZ, Jelsma JGM, van der Ploeg HP, Stijnman DPM, Huysmans MA, van der Beek AJ, van Nassau F. Barriers and facilitators influencing the implementation of the occupational health intervention 'Dynamic Work': a qualitative study. BMC Public Health. 2022 May 11;22(1):947. doi: 10.1186/s12889-022-13230-9. PMID 35546228
- [Derived] Renaud LR, Jelsma JGM, Huysmans MA, van Nassau F, Lakerveld J, Spekle EM, Bosmans JE, Stijnman DPM, Loyen A, van der Beek AJ, van der Ploeg HP. Effectiveness of the multi-component dynamic work intervention to reduce sitting time in office workers - Results from a pragmatic cluster randomised controlled trial. Appl Ergon. 2020 Apr;84:103027. doi: 10.1016/j.apergo.2019.103027. Epub 2020 Jan 10. PMID 31987512
- [Derived] Jelsma JGM, Renaud LR, Huysmans MA, Coffeng JK, Loyen A, van Nassau F, Bosmans JE, Spekle EM, van der Beek AJ, van der Ploeg HP. The Dynamic Work study: study protocol of a cluster randomized controlled trial of an occupational health intervention aimed at reducing sitting time in office workers. BMC Public Health. 2019 Feb 13;19(1):188. doi: 10.1186/s12889-019-6467-0. PMID 30760231